CLINICAL TRIAL: NCT05013827
Title: Opinions of Company Representatives About Neuromodulation for Pain: an Online Survey
Brief Title: Opinions of Company Representatives About Neuromodulation
Status: Completed | Type: Observational
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: OCEAN
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Neuromodulation; Pain; Survey
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Company representatives
  Interventions: Behavioral: Filling in an online survey

INTERVENTIONS:
Behavioral: Filling in an online survey — Company representatives are questioned about three aspects: 1) goals in treating patients with neuromodulation for pain, 2) factors that respondents expect to change according to neuromodulation for pain and 3) their definition of success of neuromodulation for pain.

SUMMARY:
The goal of this online survey is to gain further insight in the goals, expectations and definition of success for neuromodulation for pain, according to neuromodulation company representatives.

ELIGIBILITY:
Inclusion Criteria:

- Male and female adults who are involved in the management of chronic pain and more specifically in neuromodulation for pain as company representatives will be eligible to complete the survey.

Exclusion Criteria:

- Not a company representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female adults who are involved in the management of chronic pain and more specifically in neuromodulation for pain as company representatives will be eligible to complete the survey. The survey will be spread at the 2nd Joint Congress of the INS European Chapters (e-INS 2021) in Paris from 2/9/2021 to 4/9/2021.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Goals of company representatives, evaluated with a self-constructed question. | Cross-sectional evaluation during 2nd Joint Congress of the INS European Chapters (e-INS 2021) in Paris in September.
  Goals of company representatives to treat patients with neuromodulation for pain.
Company representatives expectations, evaluated with a self-constructed question. | Cross-sectional evaluation during 2nd Joint Congress of the INS European Chapters (e-INS 2021) in Paris in September.
  Factors that respondents expect to change according to neuromodulation for pain.
Company representatives definition of success of neuromodulation for pain, evaluated with a self-constructed question. | Cross-sectional evaluation during 2nd Joint Congress of the INS European Chapters (e-INS 2021) in Paris in September.
  Company representatives their definition of success of neuromodulation for pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Jette, Belgium